CLINICAL TRIAL: NCT02777411
Title: An Open-label, Dose-finding, Phase II Study to Evaluate the Safety and Immunogenicity of EV71 Vaccine in Pediatric Subjects Aged 3 to 6 Years and 6 to 35 Months Old
Brief Title: A Study to Evaluate the Safety and Immunogenicity of EV71 Vaccine in Pediatric Subjects Aged 3 to 6 Years and 6 to 35 Months Old
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Enimmune Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EV-RB1401
Record Dates: First submitted 2016-05-16; First posted 2016-05-19 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-08

CONDITIONS: Enterovirus Infections
Keywords: Vaccines; Hand, Foot and Mouth Disease; EV71 enteroviruses vaccine
MeSH Terms: conditions — Enterovirus Infections; Hand, Foot and Mouth Disease | interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Group A1 (Experimental): 3 to 6 years
  Interventions: Biological: EV71 vaccine ([0.5 μg total protein + adjuvant 150 μg AIPO4] per dose)
- Group A2 (Experimental): 3 to 6 years
  Interventions: Biological: EV71 vaccine ([1 μg total protein + adjuvant 150 μg AIPO4] per dose)
- Group A3 (Experimental): 3 to 6 years
  Interventions: Biological: EV71 vaccine ([2 μg total protein + adjuvant 150 μg AIPO4] per dose)
- Group A4 (Experimental): 3 to 6 years
  Interventions: Biological: EV71 vaccine (2 μg total protein per dose)
- Group B2 (Experimental): 6 to 35 months
  Interventions: Biological: EV71 vaccine ([0.5 μg total protein + adjuvant 150 μg AIPO4] per dose)
- Group B3 (Experimental): 6 to 35 months
  Interventions: Biological: EV71 vaccine ([1 μg total protein + adjuvant 150 μg AIPO4] per dose)
- Group B4 (Experimental): 6 to 35 months
  Interventions: Biological: EV71 vaccine (1 μg total protein per dose)

INTERVENTIONS:
Biological: EV71 vaccine ([0.5 μg total protein + adjuvant 150 μg AIPO4] per dose) — Two vaccinations at 28 days apart
  Arms: Group A1
Biological: EV71 vaccine ([1 μg total protein + adjuvant 150 μg AIPO4] per dose) — Two vaccinations at 28 days apart
  Arms: Group A2
Biological: EV71 vaccine ([2 μg total protein + adjuvant 150 μg AIPO4] per dose) — Two vaccinations at 28 days apart
  Arms: Group A3
Biological: EV71 vaccine (2 μg total protein per dose) — Two vaccinations at 28 days apart
  Arms: Group A4
Biological: EV71 vaccine ([0.5 μg total protein + adjuvant 150 μg AIPO4] per dose) — Two vaccinations at 28 days apart
  Arms: Group B2
Biological: EV71 vaccine ([1 μg total protein + adjuvant 150 μg AIPO4] per dose) — Two vaccinations at 28 days apart
  Arms: Group B3
Biological: EV71 vaccine (1 μg total protein per dose) — Two vaccinations at 28 days apart
  Arms: Group B4

SUMMARY:
The objectives of this study are to evaluate the immune response and safety profiles of two injections of EV71 vaccine administrated with or without adjuvant AlPO4 at 0.5-μg, 1-μg, 2-μg and 5-μg dose (if required) in children aged 3 to 6 years old and 0.25-μg (if required), 0.5-μg, 1-μg and 2-μg (if required) in 6 to 35 months old infants/toddlers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy children aged from 3 to 6 years old (i.e. ≥ 3 years old and < 7 years old) for Part A; from 6 to 35 months old (i.e. ≥ 6 months old and < 36 months old) for Part B at the time of first vaccination.
2. Subject's guardians were able and willing to comply with study procedures and give written informed consent.
3. Subject was able and could comply with the requirements of the protocol.
4. Subject with body temperature ≤38°C.

Exclusion Criteria:

1. Subject with previous known exposure to Enterovirus 71 (EV71).
2. Subject with a history of herpangina, hand-foot-mouth disease, acute hemorrhagic conjunctivitis associated with enterovirus infection in the past 3 months.
3. Subject with gestation < 37 weeks.
4. Subject with birth weight <2.5 kg.
5. Subject with a history of hypersensitivity to vaccines, or a history of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
6. Family history of seizures or progressive neurological disease.
7. Family history of congenital or hereditary immunodeficiency.
8. Severe malnutrition or dysgenopathy.
9. Major congenital defects or serious chronic illness, including perinatal brain damage.
10. Subject diagnosed of having autoimmune disease (e.g., celiac disease, type I diabetes, lupus (SLE), juvenile dermatomyositis, scleroderma, juvenile idiopathic arthritis (JIA), immune (or idiopathic) thrombocytopenia purpura).
11. Bleeding disorder diagnosed by a doctor or significant bruising or bleeding difficulties with IM injections or blood draws.
12. Any acute infections 7 days prior to administrate the first vaccination.
13. Use of any investigational product (including drug, vaccine) within 30 days prior to vaccination or planned use during the study period.
14. Administration of any attenuated live vaccine within 7 days prior to vaccination.
15. Use of immunoglobulins or any blood products within 3 months prior to vaccination or planned use during the study period.
16. Chronic administration (defined as > 14 days) of immunosuppressants or other immunomodulators or systemic corticosteroids within 6 months prior to vaccination.
17. Under anti-tuberculosis prevention or therapy.
18. Any condition that in the opinion of the investigator may interfere with the evaluation of study objectives.

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 122 (Actual)
Dates: Start 2014-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Solicited adverse events | 7 days after each vaccination
Unsolicited adverse events | 28 days after each vaccination
The occurrence of overall adverse events (AEs) and serious adverse event (SAEs) | Day 0 to Day 196

SECONDARY OUTCOMES:
immunoglobulin G (IgG) titers induced by the EV71 vaccine ( determined by ELISA) | Day 28, Day 56, Day 196
serum neutralizing antibody titers (NT) induced by the EV71 vaccine | Day 28, Day 56, Day 196
Seroconversion rate (SCR) based on neutralizing antibody titers | Day 28, Day 56, Day 196
change in the laboratory results based on hematology tests in each visit | Day 28, Day 56, Day 196
change in the laboratory results based on biochemistry tests in each visit | Day 28, Day 56, Day 196
change in heart rates at each visit (for the 3 to 6 years old group only) | Day 28, Day 56, Day 196
change in blood pressures at each visit (for the 3 to 6 years old group only) | Day 28, Day 56, Day 196

CONTACTS AND LOCATIONS:
Locations (4):
- Taiwan (4):
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: No